CLINICAL TRIAL: NCT01722942
Title: CHronic Use of Amiodarone aGAinSt Implantable Cardioverter-defibrillator Therapy for Primary Prevention of Death in Patients With Chagas Cardiomyopathy Study (CHAGASICS)
Brief Title: Amiodarone Against ICD Therapy in Chagas Cardiomyopathy for Primary Prevention of Death
Acronym: CHAGASICS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: InCor Heart Institute (Other)
Collaborators: Ministry of Health, Brazil (Other Government); Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Martino Martinelli Filho, PhD, MD, InCor Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHAGASICS
Record Dates: First submitted 2012-11-01; First posted 2012-11-07 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Chagas Cardiomyopathy; Non-sustained Ventricular Tachycardia; At Least 10 Points in Rassi Risk Score for Death
Keywords: Chagas cardiomyopathy; sudden cardiac death; primary prevention of death; amiodarone; implantable cardioverter defibrillator
MeSH Terms: conditions — Chagas Cardiomyopathy; Death, Sudden, Cardiac | interventions — Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ICD group (Active Comparator): ICD implantation will be performed according to the Institution protocol of each participating center; single-chamber devices are preferred and programming should prioritize the patient's own pace, avoiding ventricular stimulation.
  Interventions: Procedure: ICD implantation
- Amiodarone Group (Active Comparator): Patients randomized for this group will receive amiodarone hydrochloride (once a day) according to the following regimen:
  * Initial oral loading dose of 600 mg/day for 10 days on an outpatient basis;
  * After the loading period, an oral dose between 200 and 400 mg/day should be maintained until study termination. The determination of the optimal maintenance dose will be left at the discretion of each investigator; this dose may be based on the therapeutic response on 24-hour Holter monitoring, resting heart rate (HR), side effects, prolonged corrected QT interval (QTc), etc. Dose adjustments will be allowed throughout the study period provided the maintenance dose is kept between 200 and 400 mg/day. If the patient cannot tolerate the minimum 200 mg/day dose, amiodarone should be discontinued permanently and treatment should be considered interrupted.
  Interventions: Drug: amiodarone hydrochloride

INTERVENTIONS:
Procedure: ICD implantation — ventricular ICD implantation
  Other Names: ICD
  Arms: ICD group
Drug: amiodarone hydrochloride — amiodarone prescription
  Other Names: amiodarone
  Arms: Amiodarone Group

SUMMARY:
The primary objective is to compare the efficacy of the treatment using implantable cardioverter defibrillator (ICD) implantation to that of the treatment using amiodarone in the primary prevention of all-cause mortality in high-risk patients with Chagas cardiomyopathy and non-sustained ventricular tachycardia (NSVT).

DETAILED DESCRIPTION:
Chagas disease is an endemic problem in Latin America, where millions of people are chronically infected by Trypanosoma cruzi. The disease has also recently become clinically and epidemiologically relevant in several other countries due to social factors related to individuals migration and globalization. Chagas cardiomyopathy occurs in 30%-50% of the infected individuals, leading to considerable morbidity and mortality rates. Sudden cardiac death is the major cause of death in patients with Chagas cardiomyopathy. While implantable cardioverter defibrillator and treatment with amiodarone have been recommended and performed empirically for the secondary prevention in patients with Chagas cardiomyopathy, no consistent scientific evidence exists on the role of these therapeutic strategies for the primary prevention of Sudden cardiac death in patients with Chagas cardiomyopathy and high mortality risk.

The main hypothesis of this study is that implantable cardioverter defibrillator implantation is more efficient in the primary prevention of death in Chagas cardiomyopathy than drug therapy with amiodarone in patients with documented non-sustained ventricular tachycardia.

We should point out that the death risk will be assessed using the Rassi risk score for death prediction validated based on non-invasive variables and, depending on the results of this study, it may guide the indication of implantable cardioverter defibrillator in Chagas cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to randomization and any study procedure;
* Both genders, age > 18 years and < 75 years;
* Recent (previous 6 months) documented positive serologic test for Chagas disease in at least two different tests (indirect hemagglutination, indirect immunofluorescence, or ELISA);
* Presence of at least 10 points in Rassi risk score for death prediction;
* Presence of at least 1 episode of NSVT on Holter monitoring, defined as > 3 successive beats and duration < 30 seconds, with HR > 120 bpm is mandatory.

Exclusion Criteria:

* Participation in another study currently or < 1 year ago, except for totally unrelated observational studies;
* Other concomitant cardiovascular disease, including uncontrolled diabetes mellitus (systemic hypertension without target-organ impairment is allowed);
* Renal dysfunction (serum creatinine > 1.5 mg/dL or glomerular filtration rate (GFR) < 60 mL/min/1.73m2) or liver dysfunction with diagnosis of cirrhosis or portal hypertension or elevated serum enzymes (AST or ALT) > 3 x the upper normal limit;
* Moderate or severe chronic obstructive pulmonary disease;
* Peripheral polyneuropathy;
* Hypo or hyper-thyroidism;
* Current alcoholism or quit for <2 years;
* Mental disorder or illicit drug addiction;
* Life expectancy < 1 year, because of the disease itself or of comorbidities (including NYHA class IV CHF);
* Pregnancy or breastfeeding;
* Childbearing potential during the study (non-menopausal patients who have not undergone a safe and permanent birth control method);
* Other contraindications for the use of amiodarone: previous intolerance to the drug; HR < 55bpm; sinus node disease; type II Mobitz; fixed 2:1 AV block; advanced degree atrioventricular block (AV) block; Complete AV block; QTc > 500mseg;
* Formal indication for the use of amiodarone or defibrillator (NSVT and very disturbing palpitations, presyncope or syncope; SVT; recovery from cardiac arrest);
* Use of amiodarone in the past 6 months, except if started for < 2 weeks and if loading dose had been <10g and maintenance dose ≤100mg/day;
* Current use of betablocker considered clinically indispensable, with bradycardia < 55/min or AV block ≥ 1st degree, without pacemaker implantation;
* Current use of other medications with contraindication to the concomitant use of amiodarone;
* Persistent or permanent atrial fibrillation;
* Previous withdrawal from this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2014-10-06 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | three and half years
  All cause mortality

SECONDARY OUTCOMES:
Cardiac mortality | three and half years
  cardiac mortality
Sudden cardiac death | three and half years
  Sudden cardiac death
Worsening heart failure warranting hospitalization | three and half years
  Worsening heart failure warranting hospitalization
Need for cardiac stimulation in the ICD arm | three and half years
  Need for cardiac stimulation in the ICD arm
Need for pacemaker implantation in the amiodarone therapy arm | three and half years
  Need for pacemaker implantation in the amiodarone therapy arm

OTHER OUTCOMES:
Subgroup analyses will include gender, age ≥ or < 60 years, occurrence or not of atrial fibrillation, New York Heart Association (NYHA) functional class I and II versus III and IV, as well as Rassi score points. | three and half years
  Subgroup analyses will include gender, age ≥ or < 60 years, occurrence or not of atrial

CONTACTS AND LOCATIONS:
Overall Officials: Martino Martinelli, Prof., Principal Investigator — InCor Heart Institute
Locations (20):
- Brazil (20):
  - Hospital Universitário Walter Cantideo, Fortaleza, Ceará
  - Hospital Ana Nery, Salvador, Estado de Bahia
  - Instituto de Cardiologia do Distrito Federal, Brasília, Federal District
  - Anis Rassi Hospital, Goiânia, Goiás
  - Hospital das Clínicas de Goiania, Goiânia, Goiás
  - Santa Casa de Goiania, Goiânia, Goiás
  - Hospital Felício Rocho, Belo Horizonte, Minas Gerais
  - Hospital das Clínicas Samuel Libânio, Pouso Alegre, Minas Gerais
  - Hospital Escola da Universidade Federal do Triângulo Mineiro, Uberaba, Minas Gerais
  - Hospital Geral Universitário, Cuiabá, Mount
  - Hospital Santa Casa de Misericórdia de Curitiba, Curitiba, Paraná
  - Hospital Universitário Procape, Recife, Pernambuco
  - Hospital das Clínicas da UNICAMP, Campinas, São Paulo
  - Santa Casa de Ribeirão Preto, Ribeirão Preto, São Paulo
  - HC - FMUSP / Ribeirão Preto, Ribeirão Preto, São Paulo
  - Instituto de Moléstias Cardiovasculares, São José do Rio Preto, São Paulo
  - Heart Institute (InCor) - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo
  - Beneficiência Portuguesa, São Paulo, São Paulo
  - Escola Paulista de Medicina, São Paulo, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo

REFERENCES:
- [Derived] Martinelli-Filho M, Marin-Neto JA, Scanavacca MI, de Paola AAV, Medeiros PTJ, Owen R, Pocock SJ, de Siqueira SF; CHAGASICS investigators. Amiodarone or Implantable Cardioverter-Defibrillator in Chagas Cardiomyopathy: The CHAGASICS Randomized Clinical Trial. JAMA Cardiol. 2024 Dec 1;9(12):1073-1081. doi: 10.1001/jamacardio.2024.3169. PMID 39356542
- [Derived] Martinelli M, Rassi A Jr, Marin-Neto JA, de Paola AA, Berwanger O, Scanavacca MI, Kalil R, de Siqueira SF. CHronic use of Amiodarone aGAinSt Implantable cardioverter-defibrillator therapy for primary prevention of death in patients with Chagas cardiomyopathy Study: rationale and design of a randomized clinical trial. Am Heart J. 2013 Dec;166(6):976-982.e4. doi: 10.1016/j.ahj.2013.08.027. Epub 2013 Oct 11. PMID 24268211